CLINICAL TRIAL: NCT00184665
Title: 2 Year Efficiency and Safety Comparison of Insulin Detemir and NPH Insulin in Type 1 Diabetes.
Brief Title: Comparison of Insulin Detemir With NPH Insulin in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1595
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH
Drug: insulin aspart

SUMMARY:
This trial is conducted in Africa, Asia, Europe, Oceania, and South America. The aim of this research study is to compare the efficacy (reduction in HbA1c and in blood glucose levels) of insulin detemir compared to NPH insulin administered as basal insulin for the treatment of type 1 diabetes and to verify the safety of use (number and severity of episodes of hypoglycemia, body weight, and insulin antibodies and side effects).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Currently on basal-bolus regimen
* BMI = 35.0 kg/m2
* HbA1c =11.0%

Exclusion Criteria:

* Proliferative retinopathy or maculopathy
* Recurrent major hypoglycaemia
* Cardial problems
* Uncontrolled hypertension
* Impaired hepatic or renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2004-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
HbA1c | after a two-year trial period

SECONDARY OUTCOMES:
Adverse events
Body weight
Antibodies
Body composition
Blood glucose
Hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (27):
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Ciudad Autonoma de Bs As
  - Novo Nordisk Investigational Site, Ciudad Autónoma de BsAs
  - Novo Nordisk Investigational Site, Mar del Plata
- Australia (7):
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Hobart, Tasmania
  - Novo Nordisk Investigational Site, Melbourne, Victoria
  - Novo Nordisk Investigational Site, Darlinghurst
  - Novo Nordisk Investigational Site, Melbourne
  - Novo Nordisk Investigational Site, Stones Corner
  - Novo Nordisk Investigational Site, Woodville
- Bulgaria (2):
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Sofia
- Novo Nordisk Investigational Site, Zagreb, Croatia
- India (4):
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Chennai
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Mumbai
- Malaysia (2):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Novo Nordisk Investigational Site, Bucharest, Romania
- South Africa (3):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Bloemfontein
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, Istanbul

REFERENCES:
- [Result] Bartley PC, Bogoev M, Larsen J, Philotheou A. Long-term efficacy and safety of insulin detemir compared to Neutral Protamine Hagedorn insulin in patients with Type 1 diabetes using a treat-to-target basal-bolus regimen with insulin aspart at meals: a 2-year, randomized, controlled trial. Diabet Med. 2008 Apr;25(4):442-9. doi: 10.1111/j.1464-5491.2007.02407.x. PMID 18387078
- [Result] Gschwend MH, Aagren M, Valentine WJ. Cost-effectiveness of insulin detemir compared with neutral protamine Hagedorn insulin in patients with type 1 diabetes using a basal-bolus regimen in five European countries. J Med Econ. 2009 Jun;12(2):114-23. doi: 10.3111/13696990903080344. PMID 19545216
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com